CLINICAL TRIAL: NCT00825526
Title: HARMONY Study (Hypertension Analysis of Stress Reduction Using Mindfulness Meditation and Yoga)
Acronym: HARMONY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Sheldon Tobe, Medical Doctor, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NA 6349
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Hypertension
Keywords: Mindfulness Based Stress Reduction (MBSR); Stress Reduction; hypertension; high blood pressure; ambulatory blood pressure monitoring
MeSH Terms: conditions — Hypertension | interventions — Mindfulness-Based Stress Reduction; Therapeutics; Mindfulness

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Intervention, MBSR therapy (Experimental): Group that receives Mindfulness Based Stress Reduction Therapy immediately after randomization
  Interventions: Behavioral: Mindfulness Based Stress Reduction (MBSR) Therapy
- Delayed Treatment Arm, MBSR Therapy (Active Comparator): Group that receives Mindfulness Based Stress Reduction Therapy within 3 months of randomization
  Interventions: Behavioral: Mindfulness Based Stress Reduction (MBSR) Therapy

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction (MBSR) Therapy — The objectives of MBSR therapy are to 1) understand their personal response to stress and 2) develop techniques to change the way these patients respond and cope with stress
  Other Names: stress reduction therapy; Jon Kabat-Zinn; mindfulness meditation

SUMMARY:
The purpose of this study is to determine if Mindfulness Based Stress Reduction (MBSR) is an effective intervention for lowering blood pressure in early unmedicated hypertensives.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 to 75 years
2. Hypertension by ABPM at baseline (daytime > 135/85 mmHg or 24-hour ABPM > 130/80 mmHg)

Exclusion Criteria:

1. Use of antihypertensive within 6 months of the screening ABPM.
2. Screening office BP > 180/100 and ABPM > 160/100 mmHg.
3. Diabetes
4. Secondary hypertension
5. Renal disease (GFR < 60 ml/min or overt nephropathy)
6. History of heart attack
7. Stroke or TIA or
8. Re-vascularization procedure.
9. Active malignant disease (except non-melanoma skin cancer)
10. Epileptic seizure 6 months before the screening visit.
11. Congestive heart failure
12. Severe liver disease
13. Pregnancy or lactation period
14. Participation in a clinical trial or receipt of investigational compound or treatment in the 3 months prior to the initial screening visit.
15. Planned elective surgery during the study period except for cataract surgery

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-07; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the difference in 24-hour systolic and diastolic blood pressure between the treatment and wait-list group for the 12-week primary assessment period. | 12 weeks

SECONDARY OUTCOMES:
Changes in 24 hour ambulatory systolic and diastolic blood pressure at the end of the treatment assessment period compared to the beginning. | 12 weeks
Between and within group comparisons of MBSR on blood pressure at different times of the day including daytime, night time and work time. | 24 weeks
The proportion of patients achieving blood pressure targets (24-hour ABPM<130/80 mmHg, daytime ABPM<135/85 mmHg) at the end of the Primary Outcome period | 24 weeks
The effect of MBSR on ambulatory blood pressure by gender | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Tobe, MD, FRCP(C), Principal Investigator — Sunnybrook Health Science Centre; Brian Baker, ChB, MB, Study Chair — University Health Network, Toronto; Jane Irvine, D.Phil., C. Psych., Study Chair — York University; Susan Abbey, MD, FRCP(C), Study Chair — University Health Network, Toronto; Beth Abramson, MD, FRCPC, FACC, Study Chair — Unity Health Toronto; Martin Myers, MD, FRCPC, Study Chair — Sunnybrook Health Science Centre
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario

REFERENCES:
- [Derived] Blom K, Baker B, How M, Dai M, Irvine J, Abbey S, Abramson BL, Myers MG, Kiss A, Perkins NJ, Tobe SW. Hypertension analysis of stress reduction using mindfulness meditation and yoga: results from the HARMONY randomized controlled trial. Am J Hypertens. 2014 Jan;27(1):122-9. doi: 10.1093/ajh/hpt134. Epub 2013 Sep 14. PMID 24038797
- [Derived] Blom K, How M, Dai M, Baker B, Irvine J, Abbey S, Abramson BL, Myers M, Perkins N, Tobe SW. Hypertension Analysis of stress Reduction using Mindfulness meditatiON and Yoga (The HARMONY Study): study protocol of a randomised control trial. BMJ Open. 2012 Mar 5;2(2):e000848. doi: 10.1136/bmjopen-2012-000848. Print 2012. PMID 22396225
- See also: Overview of MBSR program — http://www.umassmed.edu/cfm/index.aspx